CLINICAL TRIAL: NCT06323720
Title: Are Signs of Central Sensitization Present in Tension-type Headache?
Brief Title: Signs of Central Sensitization in Tension-type Headache
Acronym: CSTTH
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0442
Record Dates: First submitted 2024-02-14; First posted 2024-03-21 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-02

CONDITIONS: Tension-Type Headache
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Episodic tension-type headache: Patients with 1 - 14 days of TTH/month.
  Interventions: Other: Quantitative Sensory Testing
- Chronic tension-type headache: Patients with more than 14 days TTH/month
  Interventions: Other: Quantitative Sensory Testing
- Healthy controls: Participants without tension-type headache
  Interventions: Other: Quantitative Sensory Testing

INTERVENTIONS:
Other: Quantitative Sensory Testing — Assessment of the heat and cold pain thresholds, temporal summation, conditioned pain modulation, pressure pain thresholds, electrical pain thresholds, and withdrawal reflex.

SUMMARY:
The goal of this observational study is to assess the pain sensitivity in tension-type headache patients. The main question it aims to answer is:

- Are signs of central sensitization present in tension-type headache?

Participants will be asked to fill out baseline questionnaires and they will be assessed during 1 test moment (static and dynamic quantitative sensory testing).

Researchers will compare tension-type headache patients with healthy controls to see if signs of central sensitization are only present in the tension-type headache group.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of tension headache according to globally recognized criteria (ICHD-3) or verified by a physician
2. Diagnosis of tension headache confirmed by a questionnaire (Headache Screening Questionnaire)
3. Not pregnant or given birth in the past year since a change in hormone levels can affect pain experience
4. Adults between the ages of 18 and 65
5. Proficient in the Dutch language

Exclusion Criteria:

1. Other diagnosis of headache or a mixed form
2. Other existing condition involving central nervous system sensitivity
3. Other structural neurological syndromes
4. Any condition involving the brain in the past
5. Procedure on the head, neck, or shoulder in the past 3 years
6. Currently suffering from a psychiatric condition
7. Athletes competing at a competitive level
8. Not proficient in the Dutch language
9. Currently pregnant.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will involve participation from various populations, specifically patients with episodic tension headache, patients with chronic tension headache, and healthy pain-free controls.
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pain sensitivity for heat stimuli | Baseline
  Hypersensitivity for heat pain. The heat stimulus will be delivered with the TSA-2, using a thermode.
Pain sensitivity for cold stimuli | Baseline
  Hypersensitivity for cold pain. the cold stimulus will be delivered with the TSA-2, using a thermode.
Pain sensitivity for electrical stimuli | Baseline
  Hypersensitivity for electrical pain. The electrical stimulus will be given with the Digitimer, using an electrode.
Pain sensitivity for pressure | Baseline
  Hypersensitivity for pressure pain. Pressure will be delivered using a digital algometer.
Function of the pain facilitating pathways | Baseline
  Temporal summation will be measured. This gives an idea of the (dys)function of the endogenous pain facilitation system.
Function of the pain inhibiting pathways | Baseline
  Conditioned pain modulation will be measured. This gives an idea of the (dys)function of the endogenous pain inhibiting system. A noxious conditioning heat stimulus will be given at the tibial anterior muscle. A test heat or pressure stimulus will be given at the temporalis muscle. The pain-inhibits-pain paradigm will be tested.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Van Oosterwijck, Prof, Principal Investigator — Revalidatiewetenschappen en kinesitherapie
Locations (1):
- Ghent University, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided